CLINICAL TRIAL: NCT05409235
Title: OTT166-201 A Phase 2 Randomized, Double-Masked, Vehicle-Controlled, Multicenter Study to Evaluate the Safety and Efficacy of OTT166 Ophthalmic Solution in the Treatment of Diabetic Retinopathy (DR)
Brief Title: Nesvategrast (OTT166) in Diabetic Retinopathy (DR)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: OcuTerra Therapeutics, Inc. (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OTT166-201
Record Dates: First submitted 2022-06-03; First posted 2022-06-08 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-07

CONDITIONS: Diabetic Retinopathy
Keywords: Diabetic Retinopathy; Ophthalmic solution; Non-proliferative diabetic retinopathy; Proliferative diabetic retinopathy
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- OTT166 Cohort 1 (Experimental): Participants will receive OTT166 5% twice a day (BID) for 24 weeks
  Interventions: Drug: OTT166
- OTT166 Cohort 2 (Experimental): Participants will receive OTT166 5% four times a day (QID) for 24 weeks
  Interventions: Drug: OTT166
- Vehicle control Cohort 1 (Placebo Comparator): Participants will receive vehicle control BID for 24 weeks
  Interventions: Drug: Vehicle control
- Vehicle control Cohort 2 (Placebo Comparator): Participants will receive vehicle control QID for 24 weeks
  Interventions: Drug: Vehicle control

INTERVENTIONS:
Drug: OTT166 — Participants will receive OTT166 ophthalmic solution
  Other Names: nesvategrast
  Arms: OTT166 Cohort 1; OTT166 Cohort 2
Drug: Vehicle control — Participants will receive vehicle control
  Arms: Vehicle control Cohort 1; Vehicle control Cohort 2

SUMMARY:
This study will evaluate the safety and efficacy of OTT166 Ophthalmic solution in participants with Diabetic Retinopathy.

DETAILED DESCRIPTION:
This randomized, double-masked, vehicle controlled, phase 2 study will evaluate the safety and efficacy of OTT166 ophthalmic solution in participants with diabetic retinopathy and select an optimum dosing regimen for Phase 3 pivotal trials. Approximately 210 participants diagnosed with moderately severe to severe non-proliferative diabetic retinopathy (NPDR) or mild proliferative diabetic retinopathy (PDR) and who are treatment naïve (ie, no prior anti-vascular endothelial growth factor [anti-VEGF] or laser [focal, grid, pan-retinal photocoagulation (PRP)] administered) will be randomized 2:2:1:1 into the following groups: OTT166 5% twice daily (BID), OTT166 5% four times daily (QID), vehicle control BID, vehicle control QID. Randomization will be stratified by baseline Diabetic Retinopathy Severity Scale (DRSS) score (47 or 53 or 61B). Participants with PDR (DRSS score 61B) will be capped at 20% of all randomized participants. Each group will self-administer one 50-μl eye drop of study solution (frequency as assigned) for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women ≥ 18 years of age with type 1 or 2 diabetes mellitus who have moderately severe to severe NPDR [DRSS levels 47 or 53], or mild PDR [DRSS level 61] NVE < 0.5 DA in 1 + quadrants], in whom PRP and/or anti-VEGF IVT can be safely deferred for at least 6 months per the Investigator
2. BCVA ETDRS letter score in the study eye of ≥ 69 letters (approximate Snellen equivalent of 20/40 or better)
3. Normal foveal contour
4. Treatment naïve (ie, no previous anti-VEGF or steroid treatment or PRP or laser)
5. Willing and able to return for all study visits and comply with study-related procedures
6. Able to adhere to the study dosing requirements
7. Understands and signs the written Informed Consent Form

Exclusion Criteria:

1. CST of > 325 μm

   a. Fluid in the central subfield is allowed so long as CST is ≤325 μm and there is a normal foveal contour as determined by the Central Reading Center
2. Any prior focal or grid laser photocoagulation or any prior PRP in the study eye as it pertains to treatment of DME or DR (peripheral retinal hole treated with laser is allowed)
3. Eyes with DRSS score 61 with fibrous proliferations at disc or fibrous proliferations elsewhere a. DRSS score 61B with NVE only is allowed. Any sign of fibrosis proliferation is exclusionary
4. Any prior systemic anti-VEGF treatment or IVT anti-VEGF treatment in the study eye
5. Any prior intraocular steroid injection in the study eye, inclusive of Iluvien® and Retisert® a. History of Ozurdex® and triamcinolone use prior to 12 months before study enrollment is allowed
6. Current ASNV, vitreous hemorrhage, or tractional retinal detachment visible at the screening assessments in the study eye
7. Uncontrolled glaucoma or ocular hypertension in the study eye defined as an IOP > 25 mmHg regardless of concomitant treatment with IOP-lowering medications
8. Hypertension defined as systolic > 180 mmHg or > 160 mmHg on 2 consecutive measurements (during the same visit) or diastolic > 100 mmHg
9. Screening HbA1c blood test > 12.0%
10. Renal failure (stage 4 or end-stage), dialysis, or history of renal transplant
11. History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect interpretation of the results of the study or render the participant at high risk for treatment complications
12. Initiation of intensive insulin treatment (a pump or multiple daily injections) within 4 months prior to randomization or plans to do so in the next 4 months
13. Epiretinal membrane, posterior hyaloidal traction, and/or vitreomacular traction in the study eye as determined to be significant by the Investigator
14. Previous pars plana vitrectomy in the study eye
15. Any intraocular surgery in the study eye within 90 days (3 months) prior to study enrollment
16. YAG laser treatment in the study eye within 90 days prior to study enrollment
17. Concomitant use of any topical ophthalmic medications in the study eye, including dry eye or glaucoma medications, unless on a stable dose for at least 90 days prior to study enrollment and expected to stay on stable dose throughout study participation. Topical eyedrops are allowed but not within ±10 minutes of study drop application
18. Contact lens use from time of screening throughout the study
19. Central corneal changes from dry eye that are visually significant and/or Sjogren's syndrome
20. Visually significant Fuchs endothelial dystrophy or other diagnosed conditions of corneal compromise including Anterior Basement Membrane Dystrophy, or any corneal dystrophy affecting central vision (peripheral processes are not exclusionary)
21. Chronic or recurrent uveitis in the study eye
22. Ongoing ocular infection or inflammation in either eye
23. A history of cataract surgery complicated by vitreous loss in the study eye
24. Congenital eye malformations in the study eye
25. A history of penetrating ocular trauma in the study eye
26. Cognitive impairment that, in the opinion of the investigator, could compromise compliance with the requirements of the study
27. Females of childbearing potential (ie, who are not postmenopausal for at least 1 year or surgically sterile for at least 6 weeks prior to Visit 1 - Screening/Randomization) who are lactating, or who are pregnant as determined by a positive serum pregnancy test at Visit 1 -Screening/Randomization. Women of childbearing potential must agree to use acceptable methods of birth control throughout the study a. Women who are breastfeeding or who have a positive serum hCG/urine pregnancy test at the screening or BL Visit
28. Females and males of childbearing potential unwilling or unable to utilize the following acceptable methods of birth control: tubal ligation, transdermal patch, intrauterine devices/systems, oral/implantable/injectable or contraceptives, diaphragm or cervical cap with spermicide, or vasectomized partner for females; condoms with spermicidal agent and vasectomy for males; or sexual abstinence for males and females
29. Participation in any other investigational device or drug clinical research study within 12 weeks of Visit 1 - Screening/Randomization and during the duration of enrollment
30. Contraindication to the study medications or fluorescein dye
31. Other ocular pathologies that, in the investigator's opinion, would interfere with the participant's vision in the study eye
32. Ocular media of insufficient quality to obtain fundus photographs, fluorescein angiography, and OCT images in the study eye
33. Concomitant use of Semaglutide (Wegovy®, Ozempic®, Rybelsus®), Thiazolidinediones (Actos®, Avandia®), Liraglutides (Victoza®, Saxenda®), Dulaglutide (Trulicity®), or Tirzepatide (Mounjaro®) within 12 months prior to Visit 1 (allowed if a stable dose has been established for at least 1 year of use) a. Plans to start concomitant use of Semaglutide or Thiazolidinediones during the study duration is exclusionary

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2022-07-29 (Actual); Primary Completion 2023-12-29 (Actual); Study Completion 2023-12-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carl Regillo, MD, Principal Investigator — Principal Investigator
Locations (68):
- United States (67):
  - Clinical Site 123, Peoria, Arizona
  - Clinical Site 150, Phoenix, Arizona
  - Clinical Site 111, Beverly Hills, California
  - Clinical Site 113, Encino, California
  - Clinical Site 138, Fresno, California
  - Clinical Site 129, Huntington Beach, California
  - Clinical Site 121, Pasadena, California
  - Clinical Site 127, Pasadena, California
  - Clinical Site 142, Rancho Cordova, California
  - Clinical Site 116, Riverside, California
  - Clinical Site 125, Sacramento, California
  - CinCor Site 171, Torrance, California
  - Clinical Site 160, Walnut Creek, California
  - Clinical Site 157, Coral Springs, Florida
  - Clinical Site 106, Fort Lauderdale, Florida
  - Clinical Site 131, Jacksonville, Florida
  - Clinical Site 110, Miami, Florida
  - Clinical Site 153, St. Petersburg, Florida
  - Clinical Site 117, Winter Haven, Florida
  - Clinical Site 112, ‘Aiea, Hawaii
  - Clinical Site 146, Oak Forest, Illinois
  - Clinical Site 128, Springfield, Illinois
  - Clinical Site 154, Indianapolis, Indiana
  - Clinical Site 139, Lenexa, Kansas
  - Clinical Site 166, Louisville, Kentucky
  - Clinical Site 167, Metairie, Louisiana
  - Clinical Site 163, Baltimore, Maryland
  - Clinical Site 145, Baltimore, Maryland
  - Clinical Site 103, Hagerstown, Maryland
  - Clinical Site 151, Boston, Massachusetts
  - Clinical Site 104, Boston, Massachusetts
  - Clinical Site 141, Detroit, Michigan
  - Clinical Site 155, Southaven, Mississippi
  - Clinical Site 101, Reno, Nevada
  - Clinical Site 105, Bloomfield, New Jersey
  - Clinical Site 136, Cherry Hill, New Jersey
  - Clinical Site 114, Teaneck, New Jersey
  - Clinical Site 118, Albuquerque, New Mexico
  - Clinical Site 109, Liverpool, New York
  - Clinical Site 162, Rochester, New York
  - Clinical Site 165, Raleigh, North Carolina
  - Clinical Site 143, Beachwood, Ohio
  - Clinical Site 120, Cleveland, Ohio
  - Clinical Site 152, Dublin, Ohio
  - Clinical Site 122, Edmond, Oklahoma
  - Clinical Site 135, Portland, Oregon
  - Clinical Site 158, Springfield, Oregon
  - Clinical Site 115, Kingston, Pennsylvania
  - Clinical Site 130, Beaufort, South Carolina
  - Clinical Site 133, Rapid City, South Dakota
  - Clinical Site 168, Germantown, Tennessee
  - Clinical Site 164, Knoxville, Tennessee
  - Clinical Site 169, Memphis, Tennessee
  - Clinical Site 119, Nashville, Tennessee
  - Clinical Site 161, Austin, Texas
  - Clinical Site 102, Bellaire, Texas
  - Clinical Site 108, Bellaire, Texas
  - Clinical Site 147, Burleson, Texas
  - Clinical Site 132, Fort Worth, Texas
  - Clinical Site 156, Houston, Texas
  - Clinical Site 126, McAllen, Texas
  - Clinical Site 140, San Antonio, Texas
  - Clinical Site 137, San Antonio, Texas
  - Clinical Site 144, Texas City, Texas
  - Clinical Site 159, Lynchburg, Virginia
  - Clinical Site 149, Seattle, Washington
  - Clinical Site 148, Spokane, Washington
- Clinical Site 201, Arecibo, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- OTT166 Cohort 1: Participants will receive OTT166 low dose for 24 weeks
  OTT166: Participants will receive OTT166 5% ophthalmic solution twice a day for 24 weeks
- OTT166 Cohort 2: Participants will receive OTT166 high dose for 24 weeks
  OTT166: Participants will receive OTT166 5% ophthalmic solution four time a day for 24 weeks
- Vehicle Control Cohort 1: Participants will receive vehicle control for 24 weeks
  Vehicle control: Participants will receive vehicle control twice a day for 24 weeks
- Vehicle Control Cohort 2: Participants will receive vehicle control for 24 weeks
  Vehicle control: Participants will receive vehicle control four times a day for 24 weeks
Period: Overall Study
Arm/Group | OTT166 Cohort 1 | OTT166 Cohort 2 | Vehicle Control Cohort 1 | Vehicle Control Cohort 2
Started | 75 | 76 | 38 | 36
Completed | 70 | 65 | 34 | 30
Not Completed | 5 | 11 | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- OTT166 Cohort 1: Participants received OTT166 low dose for 24 weeks
  OTT166: Participants received OTT166 5% ophthalmic solution twice a day for 24 weeks
- OTT166 Cohort 2: Participants received OTT166 high dose for 24 weeks
  OTT166: Participants received OTT166 5% ophthalmic solution four times a day for 24 weeks
- Vehicle Control Cohort 1: Participants received vehicle control for 24 weeks
  Vehicle control: Participants received vehicle control twice a day for 24 weeks
- Vehicle Control Cohort 2: Participants received vehicle control for 24 weeks
  Vehicle control: Participants received vehicle control four times a day for 24 weeks
- Total: Total of all reporting groups
Arm/Group | OTT166 Cohort 1 | OTT166 Cohort 2 | Vehicle Control Cohort 1 | Vehicle Control Cohort 2 | Total
Number analyzed (Participants) | 75 | 76 | 38 | 36 | 225
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 54 | 57 | 25 | 28 | 164
  >=65 years | 21 | 19 | 13 | 8 | 61
Age, Continuous [Mean (Full Range); unit: years] | 56.7 [24 to 89] | 56.8 [35 to 76] | 57.7 [34 to 87] | 53.9 [25 to 74] | 56.4 [24 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 32 | 13 | 12 | 95
  Male | 37 | 44 | 25 | 24 | 130
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 4 | 2 | 3 | 2 | 11
  Black or African American | 12 | 6 | 3 | 3 | 24
  White | 55 | 66 | 31 | 30 | 182
  Other | 1 | 2 | 1 | 0 | 4
  Not reported | 3 | 0 | 0 | 1 | 4
Body mass index [Mean (Full Range); unit: kg/m^2] | 34.1 [21.0 to 61.5] | 33.4 [22.1 to 62.8] | 33.2 [20.4 to 50.9] | 34.1 [22.5 to 51.5] | 34.1 [20.4 to 62.8]
Hemoglobin a1c [Mean (Full Range); unit: % of RBCs with glycosylated hemoglobin] | 8.56 [5.8 to 12.0] | 8.50 [5.5 to 12.1] | 8.37 [5.9 to 11.3] | 8.64 [5.5 to 11.1] | 8.52 [5.5 to 12.1]
Diabetic retinopathy Severity Scale at Screening [Number; unit: participants] — The Diabetic Retinopathy Severity Scale (DRSS) is a validated 12-level measure of diabetic severity. The study includes only participants' with DRSS 47, 53, or 61B. The scale was used by the imaging core lab to assess the color fundus photographs taken at each visit for the extent of diabetic retinopathy (DR). The scale is based on the counts of abnormalities in seven specified fields of the retinal photographs. The scale ranges from 10 to 85 in discreet steps with the higher number representing more extensive disease. 47 and 53 are moderately severe to severe NPDR and 61B is mild PDR.
  participants
    DRSS 47 | 47 | 46 | 23 | 23 | 139
    DRSS 53 | 13 | 14 | 7 | 6 | 40
    DRSS 61B | 15 | 16 | 8 | 7 | 46
Best corrected visual acuity [Mean (Full Range); unit: letters] — Visual function as measured by best corrected visual acuity (BCVA), the number of letters a participant can read on an Early Treatment for Diabetic Retinopathy Study (ETDRS) eye chart. A higher number of letters reflect better visual acuity with 85 letters equating to 20/20 vision on the commonly used Snellen scale.
  letters | 82.8 [69 to 94] | 82.6 [69 to 99] | 82.9 [69 to 94] | 83.4 [70 to 99] | 82.9 [69 to 99]
Central subfield thickness (CST) [Mean (Full Range); unit: microns] — The thickness (CST) of the retina in the central subfield (CST) of the fovea as measured by Optical Coherence Tomography (OCT) imaging. The higher CST the more abnormal.
  microns | 252.18 [194.7 to 299.6] | 260.72 [185.4 to 361.1] | 262.01 [217.9 to 324.6] | 256.53 [216.2 to 301.7] | 257.42 [185.4 to 361.1]
Duration of Diabetic Retinopathy [Mean (Full Range); unit: years] — The number in years since the participant's diagnosis of DR
  years | 1.699 [0.04 to 16.47] | 1.896 [0.04 to 15.61] | 2.667 [0.06 to 25.37] | 1.166 [0.04 to 7.10] | 1.843 [0.04 to 25.37]

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Who Improved by ≥ 2 Steps From Baseline in Diabetic Retinopathy Severity Scale (DRSS) Scores
Description: To characterize the efficacy of topical OTT166 in participants with DR, the Diabetic Retinopathy Severity Scale (DRSS) was used. The DRSS ranges from 10 to 85 in 12 discrete steps with higher score representing worse DR. The DRSS values were determined by the central reading center. The data reported are the estimated percentage of participants that improved by at least 2 steps from baseline. The reported data include the use of imputation according to the primary estimand as described in the protocol.
Time Frame: At week 24
Population: All participants randomized received at least one dose of study drug which is the Intent to Treat (ITT) population for the study. As was pre-specified in the study protocol, all participants assigned to receive vehicle control are reported as a single Arm/Group, Vehicle Control Combined.
Measure: Number (90% Confidence Interval); unit: estimated improvement percentage
Groups:
- OTT166 Cohort 1: Participants received OTT166 5% twice a day for 24 weeks in the study eye
- OTT166 Cohort 2: Participants received OTT166 four times a day for 24 weeks in the study eye
- Vehicle Control Combined: The combination of the vehicle control twice a day and the vehicle control four times a day groups. Comparisons are made between the two OTT166 dose groups and the combined vehicle control.
Arm/Group | OTT166 Cohort 1 | OTT166 Cohort 2 | Vehicle Control Combined
Number analyzed (Participants) | 75 | 76 | 74
estimated improvement percentage | 12.187 [5.557 to 18.816] | 12.263 [5.297 to 19.229] | 13.311 [6.260 to 20.361]
Statistical Analysis 1: Comparison: OTT166 Cohort 1 vs Vehicle Control Combined; The study was powered to provide a 90% probability to detect a 20% difference between each treatment arm and the combined vehicle control; Test type: Superiority; p = 0.5730, Mantel Haenszel; MH test is adjusted for the randomization stratification factor (Screening DRSS score 47 or 53 or 61B); difference in percentage of participants = -1.064, 90% CI 2-sided [-10.578 to 8.449] — A single imputation (non-response) when applying composite variable strategy. MI based for missing data at Week 24, assuming MAR when applying hypothetical strategy. Kept in the analysis when applying treatment policy strategy
Statistical Analysis 2: Comparison: OTT166 Cohort 2 vs Vehicle Control Combined; Test type: Superiority; p = 0.5750, Mantel Haenszel; difference in percentage of participants = -1.152, 90% CI 2-sided [-11.178 to 8.874]

2. Secondary Outcome: Proportion of Participants That Developed Worse Than Mild PDR (DRSS 65 and Above)
Description: To determine if topical OTT166 prevented or delayed the occurrence of worse than mild PDR, DRSS of 65 and above. The higher the DRSS, the greater the risk of vision loss and thus the standard of care is to treat affected patients aggressively. The reported data include the use of imputation according to the primary estimand as described in the protocol.
Time Frame: At week 24
Population: ITT population. As was pre-specified in the study protocol, all participants assigned to receive vehicle control are reported as a single Arm/Group, Vehicle Control Combined.
Measure: Number (90% Confidence Interval); unit: estimated risk percentage
Arm/Group | OTT166 Cohort 1 | OTT166 Cohort 2 | Vehicle Control Combined
Number analyzed (Participants) | 75 | 76 | 74
estimated risk percentage | 12.467 [6.105 to 18.828] | 15.316 [8.158 to 22.473] | 9.405 [3.503 to 15.307]
Statistical Analysis 1: Comparison: OTT166 Cohort 1 vs Vehicle Control Combined; Test type: Superiority; p = 0.7276, Mantel Haenszel; difference in percentage of participants = 3.119, 90% CI 2-sided [-5.314 to 11.592]
Statistical Analysis 2: Comparison: OTT166 Cohort 2 vs Vehicle Control Combined; Test type: Superiority; p = 0.8492, Mantel Haenszel; difference in percentage of participants = 5.779, 90% CI 2-sided [-3.424 to 14.982]

3. Secondary Outcome: Proportion of Participants Who Developed ASNV
Description: To determine if topical OTT166 prevented or delayed the occurrence of anterior segment neovascularization (ASNV). Measure is the percentage of patients that developed ASNV at 24 weeks. The reported data include the use of imputation according to the primary estimand as described in the protocol.
Time Frame: At week 24
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: estimated risk percentage
Arm/Group | OTT166 Cohort 1 | OTT166 Cohort 2 | Vehicle Control Combined
Number analyzed (Participants) | 75 | 76 | 74
estimated risk percentage | 4.200 [0.285 to 8.115] | 4.487 [0.288 to 8.686] | 6.068 [1.243 to 10.892]
Statistical Analysis 1: Comparison: OTT166 Cohort 1 vs Vehicle Control Combined; Test type: Superiority; p = 0.3097, Mantel Haenszel; difference in percentage of participants = -1.863, 90% CI 2-sided [-8.036 to 4.309]
Statistical Analysis 2: Comparison: OTT166 Cohort 2 vs Vehicle Control Combined; Test type: Superiority; p = 0.3414, Mantel Haenszel; difference in percentage of participants = -1.596, 90% CI 2-sided [-8.021 to 4.829]

4. Secondary Outcome: Development of PDR Worse Than Mild (Wtm) (DRSS 65 and Above)
Description: To determine if topical OTT166 prevented or delayed the occurrence of worse than mild PDR (wtmPDR). The determination was made using Kaplan-Meier methodology. The estimated percentage that progressed to wtmPDR by Week 24 is reported. The reported data include the use of imputation according to the primary estimand as described in the protocol.
Time Frame: At week 24
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | OTT166 Cohort 1 | OTT166 Cohort 2 | Vehicle Control Combined
Number analyzed (Participants) | 75 | 76 | 74
percentage of participants | 13 [7.46 to 20.75] | 17 [10.88 to 25.82] | 16 [10.24 to 25.35]
Statistical Analysis 1: Comparison: OTT166 Cohort 1 vs Vehicle Control Combined; Test type: Superiority; p = 0.397, Log Rank; Cox Proportional Hazard = 0.899, 90% CI 2-sided [0.4378 to 1.8467]
Statistical Analysis 2: Comparison: OTT166 Cohort 2 vs Vehicle Control Combined; Test type: Superiority; p = 0.605, Log Rank; Cox Proportional Hazard = 1.113, 90% CI 2-sided [0.5596 to 2.2117]

5. Secondary Outcome: Proportion of Participants Who Developed CI-DME
Description: To determine if topical OTT166 prevented or delayed the occurrence of CI-DME. CI-DME is defined as the presence of fluid in the central subfield in participants who have no fluid at baseline or CST> 325 μm. The reported data include the use of imputation according to the primary estimand as described in the protocol.
Time Frame: At week 24
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: estimated risk percentage
Arm/Group | OTT166 Cohort 1 | OTT166 Cohort 2 | Vehicle Control Combined
Number analyzed (Participants) | 75 | 76 | 74
estimated risk percentage | 14.827 [7.787 to 21.867] | 20.513 [12.331 to 28.695] | 25.459 [16.581 to 34.338]
Statistical Analysis 1: Comparison: OTT166 Cohort 1 vs Vehicle Control Combined; Test type: Superiority; p = 0.0619, Mantel Haenszel; difference in percentage of participants = -10.622, 90% CI 2-sided [-21.972 to 0.728]
Statistical Analysis 2: Comparison: OTT166 Cohort 2 vs Vehicle Control Combined; Test type: Superiority; p = 0.2483, Mantel Haenszel; difference in percentage of participants = -4.942, 90% CI 2-sided [-16.897 to 7.013]

6. Secondary Outcome: The Development of CI-DME
Description: To determine if topical OTT166 prevented or delayed the occurrence of CI-DME. CI-DME is defined as the presence of fluid in the central subfield in participants who have no fluid at baseline or CST> 325 μm. The reported data include the use of imputation according to the primary estimand as described in the protocol. The percentages of participants that developed CI-DME at Week 24 are reported.
Time Frame: At week 24
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | OTT166 Cohort 1 | OTT166 Cohort 2 | Vehicle Control Combined
Number analyzed (Participants) | 75 | 76 | 74
percentage of participants | 21 [14.44 to 30.65] | 32 [23.93 to 42.11] | 27 [19.65 to 37.37]
Statistical Analysis 1: Comparison: OTT166 Cohort 1 vs Vehicle Control Combined; Test type: Superiority; p = 0.237, Log Rank; Cox Proportional Hazard = 0.807, 90% CI 2-sided [0.4675 to 1.3920]
Statistical Analysis 2: Comparison: OTT166 Cohort 2 vs Vehicle Control Combined; Test type: Superiority; p = 0.766, Log Rank; Cox Proportional Hazard = 1.279, 90% CI 2-sided [0.7795 to 2.0981]

7. Secondary Outcome: Proportion of Participants That Developed Visually Threatening Complications (VTC) Complications (VTC)
Description: To determine if topical OTT166 prevented or delayed the occurrence of a VTC. VTC is defined as the composite outcome of PDR and/or ASNV and/or CI-DME.
Time Frame: At Week 24
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: estimated risk percentage
Arm/Group | OTT166 Cohort 1 | OTT166 Cohort 2 | Vehicle Control Combined
Number analyzed (Participants) | 75 | 76 | 74
estimated risk percentage | 23.387 [14.990 to 31.783] | 28.829 [19.730 to 37.928] | 29.838 [20.442 to 39.233]
Statistical Analysis 1: Comparison: OTT166 Cohort 1 vs Vehicle Control Combined; Test type: Superiority; p = 0.2022, Mantel Haenszel; difference in percentage of participants = -6.389, 90% CI 2-sided [-18.994 to 6.215]
Statistical Analysis 2: Comparison: OTT166 Cohort 2 vs Vehicle Control Combined; Test type: Superiority; p = 0.4476, Mantel Haenszel; difference in percentage of participants = -1.043, 90% CI 2-sided [-14.070 to 11.984]

8. Secondary Outcome: Time to Development of PDR Worse Than Mild (DRSS 65 and Above) or CI-DME
Description: To determine if topical OTT166 prevented or delayed the occurrence of PDR worse than mild (DRSS 65 and above) or CI-DME. CI-DME is defined as the presence of fluid in the central subfield in participants who have no fluid at baseline or CST> 325 μm. Participants who experienced one or more events (worse than mild PDR and/or CI-DME), the earliest event date was selected. Participants who did not experience either event were censored at the earliest of the last available assessment. Median time to event is reported if calculable.
Time Frame: From Baseline (Day 1) up to Week 24
Population: as for outcome 2
Measure: Median (90% Confidence Interval); unit: median time to event (days)
Arm/Group | OTT166 Cohort 1 | OTT166 Cohort 2 | Vehicle Control Combined
Number analyzed (Participants) | 75 | 76 | 74
median time to event (days) | NA [NA to NA] — median and 90% confidence interval were not calculable due to an insufficient number of participants having events | NA [NA to NA] — median and 90% confidence interval were not calculable due to an insufficient number of participants having events | NA [NA to NA] — median and 90% confidence interval were not calculable due to an insufficient number of participants having events
Statistical Analysis 1: Comparison: OTT166 Cohort 1 vs Vehicle Control Combined; Test type: Superiority; p = 0.268, Log Rank — log-rank test stratified by randomization stratification factor; Hazard Ratio (HR) = 0.843, 90% CI 2-sided [0.533 to 1.334]
Statistical Analysis 2: Comparison: OTT166 Cohort 2 vs Vehicle Control Combined; Test type: Superiority; p = 0.304, Log Rank; Hazard Ratio (HR) = 1.145, 90% CI 2-sided [0.738 to 1.775]

9. Secondary Outcome: Proportion of Participants With Change in DRSS Steps at Week 24 Compared to Baseline
Description: To determine the effect of OTT166 on DRSS in participants with moderately severe to severe NPDR and mild PDR treated with topical OTT166. Change in DRSS steps is defined as DR worsening or improving by 1, 2, or ≥ 3 steps along with no change. The reported data include the use of imputation according to the primary estimand as described in the protocol.
Time Frame: At week 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | OTT166 Cohort 1 | OTT166 Cohort 2 | Vehicle Control Combined
Number analyzed (Participants) | 75 | 76 | 74
percentage of participants
  Improved by ≥3 steps | 4.0 | 1.3 | 6.8
  Improved by 2 steps | 8.0 | 7.9 | 4.1
  Improved by 1 step | 18.7 | 17.1 | 27.0
  No change | 44.0 | 36.8 | 29.7
  Worsened by 1 step | 6.7 | 5.3 | 8.1
  Worsened by 2 steps | 6.7 | 2.6 | 1.4
  Worsened by ≥3 steps | 1.3 | 5.3 | 2.7
  missing | 10.7 | 23.7 | 20.3
Statistical Analysis 1: Comparison: OTT166 Cohort 1 vs Vehicle Control Combined; Test type: Superiority; p = 0.428, odds ratio; Odds ratio and p-value are from a proportional odds model with covariates for treatment group and the randomization stratification factor; Odds Ratio (OR) = 1.102, 90% CI 2-sided [0.4573 to 2.6570]
Statistical Analysis 2: Comparison: OTT166 Cohort 2 vs Vehicle Control Combined; Test type: Superiority; p = 0.419, odds ratio; [statistical method as in outcome 9, analysis 1]; Odds Ratio (OR) = 1.119, 90% CI 2-sided [0.4500 to 2.7846]

10. Secondary Outcome: Proportion of Participants With Mild PDR at Baseline Who Regressed to NPDR
Description: To determine the effect of OTT166 on DRSS in participants with mild PDR (DRSS 61B) treated with topical OTT166. Regression of disease was defined as decrease in DRSS to 53 or lower. The reported data include the use of imputation according to the primary estimand as described in the protocol.
Time Frame: At week 24
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: estimated improvement percentage
Arm/Group | OTT166 Cohort 1 | OTT166 Cohort 2 | Vehicle Control Combined
Number analyzed (Participants) | 75 | 76 | 74
estimated improvement percentage | 4.533 [0.437 to 8.629] | 2.908 [-0.687 to 6.502] | 6.149 [1.329 to 10.968]
Statistical Analysis 1: Comparison: OTT166 Cohort 1 vs Vehicle Control Combined; Test type: Superiority; p = 0.6716, Mantel Haenszel; difference in percentage of participants = -1.544, 90% CI 2-sided [-7.260 to 4.172]
Statistical Analysis 2: Comparison: OTT166 Cohort 2 vs Vehicle Control Combined; Test type: Superiority; p = 0.8414, Mantel Haenszel; difference in percentage of participants = -3.412, 90% CI 2-sided [-9.025 to 2.200]

11. Secondary Outcome: Change From Baseline in Best Corrected Visual Acuity (BCVA)
Description: To determine the effect of OTT166 on BCVA in participants with moderately severe to severe NPDR and mild PDR. BCVA was assessed by Early Treatment Diabetic Retinopathy Study (ETDRS) letters score. A higher score represents better visual function.
Time Frame: From Baseline (Day 1) up to Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: ETDRS letters
Arm/Group | OTT166 Cohort 1 | OTT166 Cohort 2 | Vehicle Control Combined
Number analyzed (Participants) | 75 | 76 | 74
ETDRS letters | -0.5829 (1.0530) | -2.3353 (1.0647) | -0.0504 (1.0594)
Statistical Analysis 1: Comparison: OTT166 Cohort 1 vs Vehicle Control Combined; Test type: Superiority; p = 0.647, ANCOVA; Mean Difference (Net) = -0.5325, 90% CI 2-sided [-2.8478 to 1.7827]
Statistical Analysis 2: Comparison: OTT166 Cohort 2 vs Vehicle Control Combined; Test type: Superiority; p = 0.945, ANCOVA; Mean Difference (Net) = -2.2849, 90% CI 2-sided [-4.6356 to 0.0658]

12. Secondary Outcome: Proportion of Participants With Lines Gained/Lost of BCVA
Description: To determine the effect of OTT166 on BCVA in participants with moderately severe to severe NPDR and mild PDR. Proportion of participants who gained/lost lines of BCVA (± 5, 10, and 15 ETDRS letters) were assessed. The reported data include the use of imputation according to the primary estimand as described in the protocol. 5 ETDRS letters = 1 line.
Time Frame: From Baseline (Day 1) up to Week 24
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | OTT166 Cohort 1 | OTT166 Cohort 2 | Vehicle Control Combined
Number analyzed (Participants) | 75 | 76 | 74
percentage of participants
  >=15 letter gain | 0 | 0 | 1.4
  10-14 letter gain | 2.7 | 1.3 | 4.1
  5-9 letter gain | 20.0 | 9.2 | 12.2
  1-4 letter gain | 30.7 | 30.3 | 27.0
  0 letter loss or gain | 8.0 | 13.2 | 5.4
  1-4 letter loss | 21.3 | 13.2 | 23.0
  5-9 letter loss | 4.0 | 9.2 | 8.1
  10-14 letter loss | 1.3 | 2.6 | 1.4
  >=15 letter loss | 1.3 | 2.6 | 0
  missing | 10.7 | 18.4 | 17.6
Statistical Analysis 1: Comparison: OTT166 Cohort 1 vs Vehicle Control Combined; Test type: Superiority; p = 0.367, odds ratio; [statistical method as in outcome 9, analysis 1]; Odds Ratio (OR) = 1.108, 90% CI 2-sided [0.6722 to 1.8276]
Statistical Analysis 2: Comparison: OTT166 Cohort 2 vs Vehicle Control Combined; Test type: Superiority; p = 0.857, odds ratio; [statistical method as in outcome 9, analysis 1]; Odds Ratio (OR) = 0.717, 90% CI 2-sided [0.4295 to 1.1981]

13. Secondary Outcome: Area Under the Curve for BCVA (ETDRS Letters) From Baseline to Week 24
Description: To determine the effect of OTT166 on BCVA in participants with moderately severe to severe NPDR and mild PDR. BCVA was assessed by ETDRS letters score. A higher score represents better functioning. AUC from baseline to 24 weeks is calculated by the linear trapezoidal method.
Time Frame: From Baseline (Day 1) up to Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: letters*day
Arm/Group | OTT166 Cohort 1 | OTT166 Cohort 2 | Vehicle Control Combined
Number analyzed (Participants) | 75 | 76 | 74
letters*day | 1997.9673 (19.3899) | 1977.5682 (19.1258) | 1993.8143 (19.4706)
Statistical Analysis 1: Comparison: OTT166 Cohort 1 vs OTT166 Cohort 2; Test type: Superiority; p = 0.437, ANCOVA; Mean Difference (Net) = 4.1531, 90% CI 2-sided [-38.7930 to 47.0991]
Statistical Analysis 2: Comparison: OTT166 Cohort 2 vs Vehicle Control Combined; Test type: Superiority; p = 0.733, ANCOVA; Mean Difference (Net) = -16.2461, 90% CI 2-sided [-59.2538 to 26.7616]

14. Secondary Outcome: Change From Baseline in Central Subfield Thickness (CST)
Description: To determine the effect of OTT166 on CST in participants with moderately severe to severe NPDR and mild PDR. CST was measured by optical coherence tomography (OCT).
Time Frame: From Baseline (Day 1) up to Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: microns
Arm/Group | OTT166 Cohort 1 | OTT166 Cohort 2 | Vehicle Control Combined
Number analyzed (Participants) | 75 | 76 | 74
microns | 14.479 (4.0974) | 9.365 (4.1020) | 10.416 (4.1107)
Statistical Analysis 1: Comparison: OTT166 Cohort 1 vs Vehicle Control Combined; Test type: Superiority; p = 0.770, ANCOVA; Mean Difference (Net) = 4.0634, 90% CI 2-sided [-4.9712 to 13.0980]
Statistical Analysis 2: Comparison: OTT166 Cohort 2 vs Vehicle Control Combined; Test type: Superiority; p = 0.424, ANCOVA; Mean Difference (Net) = -1.0507, 90% CI 2-sided [-10.1046 to 8.0032]

15. Secondary Outcome: Area Under The Curve (AUC) for Change From Baseline in CST
Description: To determine the effect of OTT166 on CST in participants with moderately severe to severe NPDR and mild PDR. CST was measured by OCT.
Time Frame: From Baseline (Day 1) up to Week 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: microns*day
Arm/Group | OTT166 Cohort 1 | OTT166 Cohort 2 | Vehicle Control Combined
Number analyzed (Participants) | 75 | 76 | 74
microns*day | 6.308 (0.0568) | 6.296 (0.0561) | 6.287 (0.0567)
Statistical Analysis 1: Comparison: OTT166 Cohort 1 vs Vehicle Control Combined; Test type: Superiority; p = 0.606, ANCOVA; Mean Difference (Net) = 0.0205, 90% CI 2-sided [-0.1043 to 0.1452]
Statistical Analysis 2: Comparison: OTT166 Cohort 2 vs Vehicle Control Combined; Test type: Superiority; p = 0.544, ANCOVA; Mean Difference (Net) = 0.0083, 90% CI 2-sided [-0.1161 to 0.1326]

16. Secondary Outcome: Proportion of Participants Who Met the Objective Rescue Criteria
Description: To determine the effect of OTT166 on the need for rescue therapy in participants with moderately severe to severe NPDR and mild PDR.
Time Frame: From Baseline (Day 1) up to Week 24
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: estimated percentage
Arm/Group | OTT166 Cohort 1 | OTT166 Cohort 2 | Vehicle Control Combined
Number analyzed (Participants) | 75 | 76 | 74
estimated percentage | 20.000 [12.752 to 29.113] | 23.684 [15.902 to 33.071] | 21.622 [14.058 to 30.969]
Statistical Analysis 1: Comparison: OTT166 Cohort 1 vs OTT166 Cohort 2; Test type: Superiority; p = 0.406, Mantel Haenszel; difference in percentage of participants = -1.544, 90% CI 2-sided [-12.247 to 9.158]
Statistical Analysis 2: Comparison: OTT166 Cohort 2 vs Vehicle Control Combined; Test type: Superiority; p = 0.605, Mantel Haenszel; difference in percentage of participants = 1.763, 90% CI 2-sided [-9.114 to 12.640]

17. Secondary Outcome: Proportion That Met Objective Rescue Therapy Criteria by Week 24
Description: To determine the effect of OTT166 on the need for rescue therapy in participants with moderately severe to severe NPDR and mild PDR. The reported data include the use of imputation according to the primary estimand as described in the protocol.
Time Frame: From Baseline (Day 1) up to Week 24
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: estimated rescue percentage
Arm/Group | OTT166 Cohort 1 | OTT166 Cohort 2 | Vehicle Control Combined
Number analyzed (Participants) | 75 | 76 | 74
estimated rescue percentage | 20 [12.752 to 29.113] | 26.684 [15.902 to 33.071] | 21.622 [14.058 to 30.969]
Statistical Analysis 1: Comparison: OTT166 Cohort 1 vs Vehicle Control Combined; Test type: Superiority; p = 0.404, Log Rank; Hazard Ratio (HR) = 0.916, 90% CI 2-sided [0.5068 to 1.6556]
Statistical Analysis 2: Comparison: OTT166 Cohort 2 vs Vehicle Control Combined; Test type: Superiority; p = 0.624, Log Rank; Hazard Ratio (HR) = 1.128, 90% CI 2-sided [0.6399 to 1.9868]

18. Secondary Outcome: Percentages of Participants at Week 24 That Had Had Rescue Therapy Administered
Description: To determine the impact of treatment with OTT166 on the time to receiving rescue therapy. Analysis was performed using the Kaplan-Meier methodology. The reported data include the use of imputation according to the primary estimand as described in the protocol. The data reported are the estimated percentages of participants at Week 24 that had had rescue therapy administered.
Time Frame: 24 Weeks
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: estimated percentage of participants
Arm/Group | OTT166 Cohort 1 | OTT166 Cohort 2 | Vehicle Control Combined
Number analyzed (Participants) | 75 | 76 | 74
estimated percentage of participants | 4 [1.67 to 10.67] | 6 [2.72 to 13.33] | 4 [1.71 to 10.87]
Statistical Analysis 1: Comparison: OTT166 Cohort 1 vs Vehicle Control Combined; Test type: Superiority; p = 0.478, Log Rank; Comparisons are made using the log-rank test stratified by randomization stratification factor; Hazard Ratio (HR) = 0.947, 90% CI 2-sided [0.2473 to 3.6295]
Statistical Analysis 2: Comparison: OTT166 Cohort 2 vs Vehicle Control Combined; Test type: Superiority; p = 0.631, Log Rank; Comparisons are made using the log-rank test stratified by randomization stratification factor; Hazard Ratio (HR) = 1.296, 90% CI 2-sided [0.3688 to 4.5512]

19. Other Pre Specified Outcome: Proportion of Participants That Develop a VTC by Week 24 for DRSS Levels 47 and 53 at Baseline
Description: A pre-specified sub group analysis of the NPDR population (DRSS 47 or 53) for the development of a VTC defined as worse than mild PDR, CI-DME or ASNV. The reported data include the use of imputation according to the primary estimand as described in the protocol.
Time Frame: 24 weeks
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: estimated risk percentage
Arm/Group | OTT166 Cohort 1 | OTT166 Cohort 2 | Vehicle Control Combined
Number analyzed (Participants) | 60 | 60 | 59
estimated risk percentage | 17.3559 [8.8130 to 25.8988] | 26.9180 [17.0207 to 36.8154] | 30.5254 [19.9191 to 41.1318]
Statistical Analysis 1: Comparison: OTT166 Cohort 1 vs Vehicle Control Combined; Test type: Superiority; p = 0.0450, Mantel Haenszel; difference in percentage of participants = -13.7727, 90% CI 2-sided [-27.1319 to -0.4134]
Statistical Analysis 2: Comparison: OTT166 Cohort 2 vs Vehicle Control Combined; Test type: Superiority; p = 0.3304, Mantel Haenszel; difference in percentage of participants = -3.8234, 90% CI 2-sided [-18.1549 to 10.5081]

20. Other Pre Specified Outcome: Proportion of Participants Who Developed CI-DME at Week 24 for Randomization Strata DRSS 47 and 53
Description: A measure of the ability to prevent CI-DME in participants with NPDR treated with OTT166. The proportion of patients that develop CI-DME (defined as new fluid in patients with no fluid at baseline or CST > 325 microns) by week 24. This is a pre-specified sub group analysis and excludes the participants in the DRSS 61B stratum. The reported data include the use of imputation according to the primary estimand as described in the protocol.
Time Frame: 24 weeks
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: estimated percentage of participants
Arm/Group | OTT166 Cohort 1 | OTT166 Cohort 2 | Vehicle Control Combined
Number analyzed (Participants) | 60 | 60 | 59
estimated percentage of participants | 13.6949 [5.9131 to 21.4767] | 20.8033 [11.7263 to 29.8803] | 28.0508 [17.7603 to 38.3414]
Statistical Analysis 1: Comparison: OTT166 Cohort 1 vs Vehicle Control Combined; Test type: Superiority; p = 0.0275, Mantel Haenszel; difference in percentage of participants = -14.8877, 90% CI 2-sided [-27.6462 to -2.1293]
Statistical Analysis 2: Comparison: OTT166 Cohort 2 vs Vehicle Control Combined; Test type: Superiority; p = 0.1790, Mantel Haenszel; difference in percentage of participants = -7.5535, 90% CI 2-sided [-21.0688 to 5.9617]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over 6 months
Groups:
- Vehicle Control Cohort 1: Participants received vehicle control twice a day for 24 weeks in the study eye
- Vehicle Control Cohort 2: Participants received vehicle control four times a day for 24 weeks in the study eye
Arm/Group | OTT166 Cohort 1 | OTT166 Cohort 2 | Vehicle Control Cohort 1 | Vehicle Control Cohort 2
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/76 | 0/38 | 0/36
Serious Adverse Events (participants affected / at risk) | 6/75 | 6/76 | 1/38 | 5/36
Other Adverse Events (participants affected / at risk) | 36/75 | 35/76 | 13/38 | 17/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OTT166 Cohort 1 (N=75) | OTT166 Cohort 2 (N=76) | Vehicle Control Cohort 1 (N=38) | Vehicle Control Cohort 2 (N=36)
Escherichia urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Accelerated hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1
Hypertensive emergency (Vascular disorders) | 0 | 0 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Cranial nerve paralysis (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 1 | 1
Alcohol abuse (Psychiatric disorders) | 1 | 0 | 0 | 0
Macular hole (Eye disorders) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OTT166 Cohort 1 (N=75) | OTT166 Cohort 2 (N=76) | Vehicle Control Cohort 1 (N=38) | Vehicle Control Cohort 2 (N=36)
Punctate keratitis (Eye disorders) | 10 | 12 | 3 | 3
Diabetic retinopathy (Eye disorders) | 5 | 3 | 3 | 3
Cataract (Eye disorders) | 3 | 4 | 0 | 1
Diabetic retinal oedema (Eye disorders) | 4 | 3 | 2 | 1
Retinal neovascularisation (Eye disorders) | 4 | 3 | 3 | 1
Dry eye (Eye disorders) | 1 | 4 | 0 | 0
Macular oedema (Eye disorders) | 0 | 0 | 2 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 2
Dysgeusia (Nervous system disorders) | 2 | 5 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 2
Hypertension (Vascular disorders) | 6 | 1 | 0 | 4

LIMITATIONS AND CAVEATS:
[Not specified]

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-10-10): https://cdn.clinicaltrials.gov/large-docs/35/NCT05409235/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-09): https://cdn.clinicaltrials.gov/large-docs/35/NCT05409235/SAP_001.pdf